CLINICAL TRIAL: NCT06550141
Title: A Phase 2 Trial of Emapalumab for the Prevention of CAR-T Cell Associated Toxicities
Brief Title: Emapalumab Prevention of CAR-T Cell Associated Toxicities
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Marcela V. Maus, M.D.,Ph.D. (Other)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor-Investigator, Marcela V. Maus, M.D.,Ph.D., Sponsor-Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-317
Record Dates: First submitted 2024-08-05; First posted 2024-08-12 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Large B-cell Lymphoma; Relapsed Non-Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma; Diffuse Large B Cell Lymphoma; Primary Mediastinal Large B-cell Lymphoma; High-grade B-cell Lymphoma; Follicular Lymphoma
Keywords: Second Line Large B-cell Non-Hodgkin's Lymphoma; Third Line Large B-cell Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — Emapalumab; Antibodies, Monoclonal; Cyclophosphamide; fludarabine phosphate; axicabtagene ciloleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Emapalumab (Experimental): Leukapheresis will happen within approximately 5 days of eligibility confirmation.
  Emapalumab is given as a single dose on Day -1 by intravenous infusion over about 1 hour.
  Lymphodepleting Chemotherapy with cyclophosphamide and fludarabine will occur once a day for 3 days (Days -5 through Day -3) by intravenous infusion over about 2-4 hours.
  Axicabtagene ciloleucel will be given once on Day 0 by intravenous infusion over about 30 minutes.
  Interventions: Drug: Emapalumab; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Drug: Axicabtagene Ciloleucel

INTERVENTIONS:
Drug: Emapalumab — An interferon gamma (IFNγ) blocking antibody
  Other Names: Human anti-interferon gamma (IFNγ) monoclonal antibody; Gamifant
Drug: Cyclophosphamide — Alkylating agent
Drug: Fludarabine Phosphate — Purine antagonist antimetabolite
Drug: Axicabtagene Ciloleucel — Autologous treatment

SUMMARY:
This research study involves assessing the impact of emapalumab as preventative management of CAR-T related cytokine release syndrome in participants with Non-Hodgkin's lymphoma (NHL).

The research study involves the following study interventions:

* Fludarabine and cyclophosphamide (Lymphodepleting Chemotherapy)
* Axicabtagene Ciloleucel
* Emapalumab

DETAILED DESCRIPTION:
This is a phase 2 multi-center, open label study that is evaluating the safety and efficacy of emapalumab in preventing toxicities associated with axicabtagene ciloleucel in subjects with second- or third-line large B-cell non-Hodgkin's lymphoma.

A phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved emapalumab for the participants specific disease, but it has been approved for other uses.

The U.S. FDA has approved axicabtagene ciloleucel for the participants specific disease.

This research study procedures include screening for eligibility, study treatment including collection of T cells (leukapheresis), lymphodepleting chemotherapy, treatment with emapalumab and axicabtagene ciloleucel, and follow-up evaluations.

Once study treatment is completed, the participants will be followed for up to 24 months.

It is expected that about 28 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with large B-cell lymphoma that is refractory to first-line chemoimmunotherapy or that relapses within 12 months of first-line chemoimmunotherapy. Or adult patients with relapsed or refractory large B-cell lymphoma after two or more lines of systemic therapy, including diffuse large B-cell lymphoma (DLBCL) not otherwise specified, primary mediastinal large B-cell lymphoma, high grade B-cell lymphoma, and DLBCL arising from follicular lymphoma.
* At least 1 measurable lesion per Lugano at time of screening.
* At least 2 weeks or 5 half-lives, whichever is shorter, must have elapsed since any prior systemic therapy at the time the subject is planned for leukapheresis, except for systemic inhibitory/stimulatory immune checkpoint therapy however steroids only require a 7-day washout.
* At least 3 half-lives must have elapsed from any prior systemic inhibitory/stimulatory immune checkpoint molecule therapy at the time the subject is planned for leukapheresis (e.g. ipilimumab, nivolumab, pembrolizumab, atezolizumab, OX40 agonists, 4-1BB agonists, etc).
* Age 18 or older
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Adequate renal, hepatic, pulmonary and cardiac function defined as:

  * ANC ≥1000/uL
  * Platelet count ≥50,000/uL
  * Absolute lymphocyte count ≥100/uL
  * Creatinine clearance (as estimated by Cockcroft Gault or CKD-EPI) ≥ 30 mL/min
  * Serum ALT/AST ≤2.5 per institutional ULN
  * Total bilirubin ≤1.5 mg/dl, except in subjects with Gilbert's syndrome.
  * Cardiac ejection fraction ≥ 40%, no clinically significant pericardial effusion, and no clinically significant ECG findings
  * Baseline oxygen saturation >92% on room air.
* Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential).
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) or follicular lymphoma unless disease free for at least 3 years.
* History of Richter's transformation of CLL.
* Autologous stem cell transplant within 6 weeks of planned axicabtagene ciloleucel infusion.
* History of allogeneic stem cell transplantation.
* Presence of uncontrolled fungal, bacterial, viral, or other infection at time of screening.
* Known history of acute or chronic active hepatitis B or C infection. Subjects with history of hepatitis infection must have cleared their infection as determined by standard serological and genetic testing per current Infectious Diseases Society of America (IDSA) guidelines.

  * Patients should also be negative for latent Tb, CMV (NAT), EBV (NAT) and adenovirus (NAT) by PCR testing.
* No evidence of active CNS disease regardless of prior CNS history.
* History or presence of CNS disorder such as seizure disorder, cerebrovascular ischemia/hemorrhage within 6 months of enrollment.
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment.
* History of symptomatic pulmonary embolism within 3 months of enrollment; ongoing anticoagulation is allowed if beyond 3 months.
* Any medical condition likely to interfere with assessment of safety or efficacy of study treatment.
* History of allergic reactions or severe immediate hypersensitivity reaction to any of the agents used in this study or compounds of similar chemical or biologic composition.
* Females who are pregnant or breastfeeding or female or male participants who are not willing to practice birth control from the time of consent through 6 months after the completion of axicabtagene ciloleucel
* In the investigators judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.
* History of autoimmune disease requiring ongoing systemic immunosuppression. Steroids are allowed up to 5mg predinosine-equivalent for adrenal insufficiency.
* Patients anticipated to require canakinumab, JAK inhibitors, TNF inhibitors, and tocilizumab for non-CAR-T management of baseline autoimmune/inflammatory disease at the time of emapalumab initiation.
* Receipt of a BCG vaccine within 12 weeks prior to Screening.
* Receipt of a live or attenuated live (other than BCG) vaccine within 4 weeks prior to screeing.
* Participants who are receiving any other investigational agents for this condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 2+ CRS per ASTCT | Day -1 to 24 months post treatment
  Assessed using American Society for Transplantation and Cellular Therapy (ASTCT). All participants will be monitored and assessed for grade 2+ cytokine release syndrome (CRS) for 24 months after post treatment.

SECONDARY OUTCOMES:
Rate and severity of ICANS as per ASTCT | 30 days
  Assessed using American Society for Transplantation and Cellular Therapy (ASTCT). The rate and severity of immune cell associated neurotoxicity syndrome (ICANS) within the first 30 days of infusion.
Objective response rate (ORR) | Day -1 to 24 months post treatment
  The incidence of either a complete response or a partial response by Lugano. All subjects that do not meet the criteria for an objective response by the analysis data cutoff date will be considered non-responders.

OTHER OUTCOMES:
Duration of response (DOR) | From First Objective Response until date of first documented disease progression or date of death from any cause, assessed up to 24 months post treatment
  Among subject who experience an objective response the date of their first objective response to disease progression per Lugano or death regardless of cause. Subjects not meeting the criteria for progression or death by the analysis data cutoff date will be censored at their last evaluable disease assessment date and their response will be noted as ongoing.
Progression-free Survival (PFS) | From Day 0 until date of first documented disease progression or date of death from any cause, assessed up to 24 months post treatment
  The time from the axicabtagene ciloleucel infusion date to the date of disease progression per Lugano or death from any cause. Subjects not meeting the criteria for progression by the analysis data cutoff date will be censored at their last evaluable disease assessment date.
Overall survival (OS) | From Day 0 until documented date of death from any cause, assessed up to 24 months post treatment
  The time from axicabtagene ciloleucel infusion to the date of death. Subjects who have not died by the analysis data cutoff date will be censored at their last contact date.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Frigault, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation